CLINICAL TRIAL: NCT01803867
Title: A Double-Blind, Placebo-Controlled, Single Ascending Intravenous Infusion Study of Recombinant Human Immunoglobulin M (rHIgM22) in Patients With Multiple Sclerosis (MS)
Brief Title: An Intravenous Infusion Study of rHIgM22 in Patients With Multiple Sclerosis
Acronym: M22
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM22-MS-1004
Record Dates: First submitted 2013-02-26; First posted 2013-03-04 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Multiple Sclerosis
Keywords: MS; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rHIgM22 (Placebo Comparator): Cohorts 1-5: In each dosing cohort, the first 2 eligible patients will be enrolled and randomized 1:1 to receive rHIgM22 or placebo, and monitored for safety for a minimum of 7 days before the remaining 8 patients in the cohort are randomized (7 active: 1 placebo) and dosed.
  Expanded Cohort: Upon establishment of a Maximally Tolerated Dose (MTD), a new group of 21 patients will be enrolled in an Expansion Cohort. Randomly assigned in a 1:1:1 ratio to 1 of 3 treatment groups: placebo, Investigational Product (IP) at MTD, or IP at one full dose level lower than MTD.
  Interventions: Drug: rHIgM22

INTERVENTIONS:
Drug: rHIgM22 — Administered via IV infusion
  Other Names: M22

SUMMARY:
This is a Phase I, multi-center, double-blind, randomized, placebo-controlled, dose-escalation study designed to evaluate safety, tolerability, pharmacokinetics, and immunogenicity of single intravenous (IV) administrations of rHIgM22 in patients with all clinical presentations of MS.

ELIGIBILITY:
Inclusion Criteria:

* Able to give written informed consent, with adequate cognitive function to sign the IRBapproved informed consent
* Meet diagnostic criteria for MS, as defined by revised (2010) McDonald criteria
* Man or woman aged 18 to 70 years, inclusive
* Women of childbearing potential must have a negative serum pregnancy test at the Screening Visit and
* Women of childbearing potential and engaged in heterosexual relations must agree to practice adequate contraception for at least 60 days after study dosing. Women of childbearing potential and not engaged in heterosexual relations or not practicing adequate contraception must agree to remain abstinent for at least 60 days after study dosing practice adequate contraception for the duration of the study
* Agree to remain in the hospital for the 48 hour post infusion observation period, and can be contacted in case of an emergency once discharged

Exclusion Criteria:

* Serum creatinine ≥1.5 mg/dL
* Aspartate aminotransferase (AST), Alanine aminotransferase (ALT) or alkaline phosphatase ≥1.5 times the upper limit of normal
* Angina, uncontrolled hypertension, clinically significant cardiac arrhythmias (including atrial fibrillation), any other clinically significant cardiovascular abnormality or clinically significant abnormal ECG
* Immune-mediated disorder other than MS that in the Investigator's judgment, may affect the interpretation of results or the patient's ability to safely complete the study
* Any clinically significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, allergic or anaphylactic reasons, or other major diseases (other than MS), that in the Investigator's judgment, may affect the interpretation of results or patient's ability to safely complete the study. This includes a suicide attempt within the past 1 year or severe suicidal ideation within the past 6 months or patients who in the opinion of the Investigator are at significant risk of suicidal behavior
* MS relapse within 30 days prior to screening or treatment with systemic (oral, IV or IM) corticosteroids, except for minimally absorbed topical or inhalational preparations, within the 30 days prior to the Screening Visit
* Initiation of interferon-beta 1b (Betaseron,a extavia), interferon beta-1a (Avonex, a Rebif a), glatiramer acetate (copaxone), natalizumab (Tysabri), or fingolimod (Gilenya), or dimethyl fumarate (Tecfidera ®) within the 90 days prior to the Screening Visit, or any change in the dosing regimen of these drugs within the 30 days prior to the Screening Visit. Initiation of teriflunomide (AUBAGIO®) or any change in the dosing regimen of this drug within 90 days prior to the Screening Visit.
* Treatment with any of the following medications within the 12 months prior to Day 1 of the study: daclizumab, azathioprine, methotrexate, IV immunoglobulin, plasmaphoresis, or mycophenolate mofetil; or discontinuation of teriflunomide (AUBAGIO®) within 12 months prior to Day 1.
* History of clinically significant infusion reactions with administration of biologics, including plasma exchange, intravenous immunoglobulin, and other monoclonal antibodies such as natalizumab (Tysabri)
* Prior treatment with total lymphoid irradiation, T cell or T-cell receptor vaccination, alemtuzumab, mitoxantrone, cyclophosphamide, or rituximab
* Received any investigational agent or therapy up to 30 days or 4 pharmacokinetic half-lives (whichever is longer) prior to Screening Visit or plans to enroll in another investigational trial at any time during this study
* Contraindication to brain MRI or inability to tolerate brain MRI

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-03; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single ascending doses of the human monoclonal rHIgM22 in patients with MS. | 90 Days
  Monitoring of adverse events (AEs) will be conducted throughout the study. Adverse events, including serious adverse events will be recorded in the case report forms (CRFs).

SECONDARY OUTCOMES:
Measure the pharmacokinetics (PK) of single ascending doses of rHIgM22 | Day 1 through Day 180
  PK parameters will include; The maximum measured plasma concentration (Cmax), time to maximum plasma concentration (Tmax), half-life (T1/2), and the area under the concentration curve from time 0 to the concentration at last time point (AUC (0-last)).
Measure the pharmacodynamics of single ascending doses of rHIgM22 using the Expanded Disability Status Scale (EDSS) | Day 1 through Day 180

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Carrazana, MD, Study Director — Acorda Therapeutics
Locations (16):
- United States (16):
  - Acorda Investigational Site, Long Beach, California
  - Acorda Investigational Site, Palo Alto, California
  - Acorda Investigational Site, Sacramento, California
  - Acorda Investigational Site, Stanford, California
  - Acorda Investigational Site, Aurora, Colorado
  - Acorda Investigational Site, Centennial, Colorado
  - Acorda Investigational Site, Indianapolis, Indiana
  - Acorda Investigational Site, Kansas City, Kansas
  - Acorda Investigational Site, Baltimore, Maryland
  - Acorda Investigational Site, St Louis, Missouri
  - Acorda Investigational Site, Rochester, New York
  - Acorda Investigational Site, Providence, Rhode Island
  - Acorda Investigational Site, Knoxville, Tennessee
  - Acorda Investigational Site, Dallas, Texas
  - Acorda Investigational Site, Burlington, Vermont
  - Acorda Investigational Site, Seattle, Washington